CLINICAL TRIAL: NCT06862024
Title: Effect of PechaKucha (PK) Presentation Method on Nursing Students' Satisfaction Level With Deep Breathing and Cough Exercise Skills and Education Method
Brief Title: Effect of PechaKucha (PK)Presentation Method on Nursing Students' Satisfaction Level With Deep Breathing and Cough Exercise Skills and Education Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Vildan Budak, Mscn, Eastern Mediterranean University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EasternEMU
Record Dates: First submitted 2025-02-22; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: PechaKucha Presentation; Traditional PowerPoint Presentation
Keywords: PechaKucha; Nursing students; breathing exercise; satisfaction,
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PK Presentation (Experimental): Giving Deep Breathing and Cough exercises with PK presentation method
  Interventions: Behavioral: Deep Breathing and Cough Exercise Skills; Behavioral: Satisfaction with the training method
- Power Point Presentation (Active Comparator): Giving Deep Breathing and Cough exercises using traditional Power Point presentation method
  Interventions: Behavioral: Deep Breathing and Cough Exercise Skills; Behavioral: Satisfaction with the training method

INTERVENTIONS:
Behavioral: Deep Breathing and Cough Exercise Skills — Ability to apply deep breathing and cough exercise skills will be examined.
Behavioral: Satisfaction with the training method — The level of satisfaction with the training provided will be determined with the PechaKucha presentation.

SUMMARY:
ABSTRACT

Aim: The aim of this study is to examine the effect of the PK presentation method on nursing students' deep breathing and cough exercise skills and the students' level of satisfaction with this method.

Design: The sample of the study consisted of students studying in the 2nd year of the Nursing Department of a foundation university and taking the Fundamentals of Nursing course (n=96). Experimental (n=48) and control (n=48) groups were determined using a randomization program. While the students in the experimental group were taught deep breathing and cough exercises with the PK presentation method, the control group was trained with a traditional Power Point presentation. As data collection tools, student information form, deep breathing and cough exercise skill checklist and Visual Analog Scale measurement tool were used to determine the level of satisfaction with the training method.

Keywords: PechaKucha, Nursing students, respiratory exercise, satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria Taking the Fundamentals of Nursing course for the first time attending the course on the day of the course

Exclusion Criteria:

* Students taking the course for the second time and those who did not attend the course on the day of the training were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Satisfaction level of Deep Breathing and Cough Exercise Skills Training given with PechaKucha presentation method | 3 day
  Visual Analog Scale A visual analog scale was used to measure students' satisfaction levels with the given training method, where students can score between 1 and 10..
Effect of PechaKucha presentation method on Deep Breathing and cough exercise skills | 3 day
  The steps of the Deep Breathing and Cough Exercise were prepared in accordance with the literature. Expert opinions were obtained for the scope validity of the prepared checklist according to the Davis technique. According to this technique, expert opinions are graded in 4 stages; 1-"Not appropriate", 2-"Item needs to be brought into appropriate form", 3-"Appropriate but minor changes are required", 4-"Very appropriate". The number of experts who gave 3 and 4 points to all items in the scale is divided by the total number of experts who received opinions and the Scope Validity Index (CVI) is obtained. In order for the items to be evaluated as sufficient in terms of scope validity, the "Scope Validity Index" must be above 0.80 [15]. In this technique, opinions are obtained from at least 3 and at most 20 experts. In this direction, expert opinions were obtained from 9 faculty members specialized in the field of Fundamentals of Nursing for the scope validity of the checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Cevheroglu, Assit. Dr., Principal Investigator — Eastern Mediterranean University; Vildan Budak, MScN, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
will be re-evaluated at the end of the study

REFERENCES:
- [Result] Haramba SJ, Millanzi WC, Seif SA. Enhancing nursing student presentation competences using Facilitatory Pecha kucha presentation pedagogy: a quasi-experimental study protocol in Tanzania. BMC Med Educ. 2023 Sep 3;23(1):628. doi: 10.1186/s12909-023-04628-z. PMID 37661279
- [Result] Haramba SJ, Millanzi WC, Seif SA. Effects of pecha kucha presentation pedagogy on nursing students' presentation skills: a quasi-experimental study in Tanzania. BMC Med Educ. 2024 Aug 31;24(1):952. doi: 10.1186/s12909-024-05920-2. PMID 39217328
- [Result] Erol Ursavas F, Tok Ozen A, Ozaras Oz G. Evaluation of the effect of stoma care training using the pechakucha method on stoma care skills and anxiety in nursing students: A single-blind randomized controlled trial. Nurse Educ Pract. 2024 Oct;80:104106. doi: 10.1016/j.nepr.2024.104106. Epub 2024 Aug 22. PMID 39191200
- [Derived] Cevheroglu S, Firat Kilic H, Budak V. The effect of the PechaKucha presentation method on nursing students' deep breathing and coughing exercise skills and their satisfaction with the educational method: a randomized controlled trial. BMC Med Educ. 2025 Dec 2;25(1):1667. doi: 10.1186/s12909-025-08258-5. PMID 41331646